CLINICAL TRIAL: NCT01214499
Title: Prospective, Controlled and Randomized Clinical Trial on Cardiac Cell Regeneration With Laser and Autologous Bone Marrow Stem Cells, in Patients With Coronary Disease and Refractory Angina
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Dr. Guillermo Reyes Copa, Cardiovascular Surgery Service, Hospital Universitario de La Princesa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMR-SC-02
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Angina; Coronary Disease
Keywords: Refractory angina; Transmyocardial revascularization; Stem cells; Diffuse coronary disease not amenable to percutaneous coronary intervention, and angina, despite proper medical treatment
MeSH Terms: conditions — Angina Pectoris; Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Control (Active Comparator): Transmyocardial revascularization (TMR) with Holmium YAG (yttrium aluminium garnet) laser, according to habitual clinical practice in the Department of Cardiovascular Surgery.
  Interventions: Procedure: Transmyocardial revascularization (TMR) with Holmium YAG laser
- Experimental Treatment (Experimental): Transmyocardial revascularization (TMR) with Holmium YAG laser plus the patient's own stem cells extracted from bone marrow.
  Interventions: Procedure: Transmyocardial revascularization (TMR) with Holmium YAG laser plus the patient's own stem cells extracted from bone marrow.

INTERVENTIONS:
Procedure: Transmyocardial revascularization (TMR) with Holmium YAG laser — Transmyocardial revascularization (TMR) is a surgical procedure that uses a laser to create channels through the myocardial, so this laser stimulates local angiogenesis and provides blood in the ischemic area.
  Arms: Treatment Control
Procedure: Transmyocardial revascularization (TMR) with Holmium YAG laser plus the patient's own stem cells extracted from bone marrow. — The system called PHOENIXTM consists of a laser probe with Holmium:YAG energy capable of creating transmural channels in the myocardium. Surrounding this fibre 3 needles with side holes are arranged so that the implantation of stem cells is done on the edges of the channel and not on the channel itself. This device is capable of distributing stem cells in those channels created by the laser, carrying out both procedures simultaneously.
  Arms: Experimental Treatment

SUMMARY:
Coronary disease is one of the most frequent pathology of the modern world and the leading cause of death in the investigators country. In Spain more than 50.000 coronary percutaneous intervention and more than 5.000 coronary artery bypass graft (CABG) procedures are performed every year. Despite this data about 12% of patients have diffuse coronary disease and are not candidates to conventional therapies. Also between 15-25% of patients undergoing coronary bypass grafting receive an incomplete revascularization due to the poor quality of the coronary vessels.

Transmyocardial revascularization (TMR) is a surgical procedure that uses a laser to create channels through the myocardial, so this laser stimulates local angiogenesis and provides blood in the ischemic area. Results of this procedure have shown clear benefits in terms of reduction of angina and increase of survival of patients, compared to medical treatment.

Cell therapy in heart disease is offering in recent years encouraging results despite the methodological difficulties that being able to use this technique sometimes involves. The basis lies in the potential ability of stem cells to differentiate into any type of adult cell. In the case of cardiac cell therapy, stem cells can differentiate into myocardial cells or vascular cells capable of developing angiogenesis. Further studies are needed to draw firm conclusions about the clinical impact that the use of stem cells has on cardiovascular disease.

Recently a system has been developed to create, at the same time and in a simple and effective way, the laser channels and the introduction of stem cells on the edges of these channels. This system called PHOENIX ™ consists of a laser probe capable of creating transmural channels in the myocardium.

Based on the what has just been explained, it is quite possible that the combination of both therapies can increase successful results regarding the reduction in angina these patients need. Initially, and after having some experience with this type of treatment, the results could be analyzed and compared with the results obtained through laser therapy, with the help of a controlled clinical trial, such as the one the investigators are proposing.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with at least one area of myocardial ischemia or chronic myocardial infarction of the left ventricle demonstrated by any imaging technique not amenable to conventional revascularization and angina refractory to medical treatment.
* Ejection fraction> 25% measured in the six months prior to the procedure.
* Participants must be mentally competent to give consent for inclusion in the clinical trial

Exclusion Criteria:

* Patients with unstable angina defined as the need for intravenous nitrates at the time of surgery.
* Recent myocardial infarction (within 15 days before the procedure).
* Patients with decompensated heart failure at the time of surgery.
* Severe or life threatening arrhythmia (ventricular tachycardia or fibrillation) in the week before the procedure.
* Patients requiring some type of concomitant valvular surgery.
* Patients with severe obstructive lung disease criteria who are considered as not capable of bearing general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
New York Heart Association (NYHA)classification for angina | one year
  The main variable under study is the percentage of patients achieving a decrease in two levels of the NYHA classification for angina.

SECONDARY OUTCOMES:
The demographic, intra and postoperative variables | one year
  The demographic variables and patients' cardiovascular history will be collected. All the intra and postoperative variables will be collected, as well as the data obtained by cytometry (amount of cells injected into each appropriate patient)
Tests | one year
  Before surgery and 12 months after it a test of ischemia provocation through isotopes will be carried out in order to measure the percentage of ischemic area (SPECT or Single Photon Emission Computed Tomography) and maximum effort capacity before the occurrence of the angina.
  The ejection fraction, the end-systolic volume and the end-diastolic volume of the left ventricle will be examined through an echocardiogram and a pre- and postoperative cardiac magnetic resonance imaging study.
Quality of Life | one year
  The EQ-5D questionnaire (standardised instrument for use as a measure of health outcome)will be completed for the subjective assessment of the quality of life that the patient perceives to have.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Reyes Copa, Physician Doctor, Principal Investigator — Cardiovascular Surgey Service, Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

REFERENCES:
- [Background] Lopez-Palop R, Moreu J, Fernandez-Vazquez F, Hernandez Antolin R. [Spanish Cardiac Catheterization and Coronary Intervention Registry. 15th official report of the Spanish Society of Cardiology Working Group on Cardiac Catheterization and Interventional Cardiology (1990-2005)]. Rev Esp Cardiol. 2006 Nov;59(11):1146-64. Spanish. PMID 17144990
- [Background] Mukherjee D, Bhatt DL, Roe MT, Patel V, Ellis SG. Direct myocardial revascularization and angiogenesis--how many patients might be eligible? Am J Cardiol. 1999 Sep 1;84(5):598-600, A8. doi: 10.1016/s0002-9149(99)00387-2. PMID 10482164
- [Background] Weintraub WS, Jones EL, Craver JM, Guyton RA. Frequency of repeat coronary bypass or coronary angioplasty after coronary artery bypass surgery using saphenous venous grafts. Am J Cardiol. 1994 Jan 15;73(2):103-12. doi: 10.1016/0002-9149(94)90198-8. PMID 8296729
- [Background] Bridges CR, Horvath KA, Nugent WC, Shahian DM, Haan CK, Shemin RJ, Allen KB, Edwards FH; Society of Thoracic Surgeons. The Society of Thoracic Surgeons practice guideline series: transmyocardial laser revascularization. Ann Thorac Surg. 2004 Apr;77(4):1494-502. doi: 10.1016/j.athoracsur.2004.01.007. PMID 15063304
- [Background] Allen KB, Dowling RD, Angell WW, Gangahar DM, Fudge TL, Richenbacher W, Selinger SL, Petracek MR, Murphy D. Transmyocardial revascularization: 5-year follow-up of a prospective, randomized multicenter trial. Ann Thorac Surg. 2004 Apr;77(4):1228-34. doi: 10.1016/j.athoracsur.2004.01.008. PMID 15063241
- [Background] Allen KB, Dowling RD, Schuch DR, Pfeffer TA, Marra S, Lefrak EA, Fudge TL, Mostovych M, Szentpetery S, Saha SP, Murphy D, Dennis H. Adjunctive transmyocardial revascularization: five-year follow-up of a prospective, randomized trial. Ann Thorac Surg. 2004 Aug;78(2):458-65; discussion 458-65. doi: 10.1016/j.athoracsur.2004.04.049. PMID 15276496
- [Background] Abdel-Latif A, Bolli R, Tleyjeh IM, Montori VM, Perin EC, Hornung CA, Zuba-Surma EK, Al-Mallah M, Dawn B. Adult bone marrow-derived cells for cardiac repair: a systematic review and meta-analysis. Arch Intern Med. 2007 May 28;167(10):989-97. doi: 10.1001/archinte.167.10.989. PMID 17533201
- [Background] Haider HKh. Bone marrow cells for cardiac regeneration and repair: current status and issues. Expert Rev Cardiovasc Ther. 2006 Jul;4(4):557-68. doi: 10.1586/14779072.4.4.557. PMID 16918274
- [Background] Haider HKh, Ashraf M. Bone marrow stem cell transplantation for cardiac repair. Am J Physiol Heart Circ Physiol. 2005 Jun;288(6):H2557-67. doi: 10.1152/ajpheart.01215.2004. PMID 15897328
- [Background] Anversa P, Leri A, Kajstura J, Nadal-Ginard B. Myocyte growth and cardiac repair. J Mol Cell Cardiol. 2002 Feb;34(2):91-105. doi: 10.1006/jmcc.2001.1506. PMID 11851350
- [Background] Klein HM, Ghodsizad A, Borowski A, Saleh A, Draganov J, Poll L, Stoldt V, Feifel N, Piecharczek C, Burchardt ER, Stockschlader M, Gams E. Autologous bone marrow-derived stem cell therapy in combination with TMLR. A novel therapeutic option for endstage coronary heart disease: report on 2 cases. Heart Surg Forum. 2004;7(5):E416-9. doi: 10.1532/HSF98.20041095. PMID 15799915
- [Background] Patel AN, Spadaccio C, Kuzman M, Park E, Fischer DW, Stice SL, Mullangi C, Toma C. Improved cell survival in infarcted myocardium using a novel combination transmyocardial laser and cell delivery system. Cell Transplant. 2007;16(9):899-905. doi: 10.3727/096368907783338253. PMID 18293888
- [Background] Reyes G, Allen KB, Aguado B, Duarte J. Bone marrow laser revascularisation for treating refractory angina due to diffuse coronary heart disease. Eur J Cardiothorac Surg. 2009 Jul;36(1):192-4. doi: 10.1016/j.ejcts.2009.03.022. Epub 2009 Apr 25. PMID 19394846
- [Background] Karch FE, Lasagna L. Toward the operational identification of adverse drug reactions. Clin Pharmacol Ther. 1977 Mar;21(3):247-54. doi: 10.1002/cpt1977213247. PMID 837643